CLINICAL TRIAL: NCT00918359
Title: Following Study: Heat Intolerance- A Lesson From Global Genomic Response in Lymphocytes
Brief Title: Heat Intolerance- A Lesson From Global Genomic Response in Lymphocytes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: heller institute, Medical Corps, Israel Defense Force
Other Study IDs: 782-2008-IDF-CTIL
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Heat Intolerance; Genotypic Variations; Gene Expression; Genomic Markers for Predisposition of Heat Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (2):
- HI: Subjects who experienced heat exhaustion or heat stroke in their past and will be identified by heat tolerance test (HTT) as Heat Intolerance .
- HT: Subjects who experienced heat exhaustion or heat stroke in their past and will be identified by heat tolerance test (HTT) as Heat Tolerance .

SUMMARY:
Heat Intolerance (HI) is a life threatening deficiency that can lead to heat exhaustion, heat stroke (and possibly death) in a large number of military and civilian occupational groups. We have demonstrated malfunction of transcriptional pathways in the heat stressed HI phenotype and an altered gene expression profile compared to Heat Tolerant (HT) individuals. Such differences are evident even under normothermic basal/comfort conditions. Heat and exercise challenges during the heat tolerance test (HTT) further emphasize the differences between the groups, particularly during recovery at comfort temperatures. Our results indicate that it may be possible to identify markers of heat intolerance. To achieve this goal, we plan to design a cellular (lymphocyte) HTT experimental model and detect gene expression profiles using customized DNA microarrays and bioinformatic tools (the genes selected will be based on our previous DNA microarray studies). Lymphocyte samples collected from HT and HI individuals under resting/comfort conditions will be examined. Treatments and analyses are designed to reveal HI-associated gene-expression profiles (constitutive or inducible), and thereby find lymphocyte markers to identify individuals predisposed to heat injury. The identification of such subjects could prevent unnecessary loss of life. Notably, the rapidly changing climate in our era increases the number of occupation/age groups in which manifestations of HI will appear.

ELIGIBILITY:
Inclusion Criteria:

* Experienced heat exhaustion or heat stroke in their past
* Participating in heat tolerance tests (HTT)

Exclusion Criteria:

* Unambiguous result of the HTT
* HTT stop by the subject decision

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Blood samples of HT and HI subjects will be collected from volunteers who experienced heat exhaustion or heat stroke in their past and participating in heat tolerance test (HTT). The test, using conservative criteria discriminates between HI and HT groups. The distinction between HI and HT groups occurs only following analyses of the HTT.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-05

CONTACTS AND LOCATIONS:
Locations (1):
- Heller Institute of Medical Research, Ramat Gan, Israel